CLINICAL TRIAL: NCT01819103
Title: Evaluation of the Methods and Management of Acute Coronary Events-4: Investigating Variation in Hospital Acute Coronary Syndrome Outcomes
Brief Title: Investigating Variation in Hospital Acute Coronary Syndrome Outcomes
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Oras Alabas, Dr, University of Leeds
Other Study IDs: 12/WM/0431
Record Dates: First submitted 2013-03-23; First posted 2013-03-27 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Mortality; Acute Myocardial Infarction; Drug Adherence; Drug Compliance; Health-related quality of life
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute myocardial infarction: Drug Adherence

SUMMARY:
To investigate the causes of hospital variation in outcomes from acute coronary syndromes in England and develop recommendations for improving patient care.

DETAILED DESCRIPTION:
Over the last few years the chance of dying from a heart attack in England and Wales has reduced dramatically. Even so, there remain huge differences in mortality between hospitals. For example, up to a third of patients with a heart attack who attend hospitals in England are more likely to die than would be expected. That is, the type of treatment and the risk of death depend upon where a patient lives and which hospital they attend. In part, the variation in death may be due to the services available at the hospital or to factors such as socioeconomic deprivation. It may also relate to other factors such as depression, cardiac rehabilitation, patient experience of hospital care and whether patients take their medication after discharge from hospital.

Notably, the challenges posed by poor drug adherence to secondary prevention medications are recognised by the World Health Organisation as the highest area of priority for improving individual health throughout the world. In addition, Patient Reported Outcome Measures (PROMs) are set to be the cornerstone of the evaluation of patient experiences of National Health Service quality of care.

Using statistical approaches that include measures of quality of life, we propose to examine data about heart attacks in England and investigate the 'postcode lottery of care'. Our aim, using regional data about heart attacks is to identify and measure the effects of hospital care. This research will identify hospital qualities that promote improved patient care. In doing so, best practice will be highlighted and healthcare policy changed so that all patients will have an equal chance of surviving a heart attack.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years, both sexes, acute admission to the acute Trust with suspected acute coronary syndrome (ACS).

Exclusion Criteria:

Patients at a terminal stage of any illness, and those in whom follow up would be inappropriate or impractical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 5555 consented patients were recruited from acute Trusts in England.
Sampling Method: Non-Probability Sample
Enrollment: 5555 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months

SECONDARY OUTCOMES:
Drug Adherence | 12 month

OTHER OUTCOMES:
Health related quality of life assessement | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Chris P Gale, PhD, Principal Investigator — University of Leeds

REFERENCES:
- [Derived] Munyombwe T, Dondo TB, Hall M, Nadarajah R, Hurdus B, Aktaa S, Haris M, Keeley A, West R, Hall A, Norman P, Gale CP. Cohort profile: Evaluation of the Methods and Management of Acute Coronary Events (EMMACE) Longitudinal Cohort. Eur Heart J Qual Care Clin Outcomes. 2023 Aug 7;9(5):442-446. doi: 10.1093/ehjqcco/qcad040. PMID 37451698
- [Derived] Dondo TB, Munyombwe T, Hall M, Hurdus B, Soloveva A, Oliver G, Aktaa S, West RM, Hall AS, Gale CP. Sex differences in health-related quality of life trajectories following myocardial infarction: national longitudinal cohort study. BMJ Open. 2022 Nov 8;12(11):e062508. doi: 10.1136/bmjopen-2022-062508. PMID 36351712
- [Derived] Munyombwe T, Dondo TB, Aktaa S, Wilkinson C, Hall M, Hurdus B, Oliver G, West RM, Hall AS, Gale CP. Association of multimorbidity and changes in health-related quality of life following myocardial infarction: a UK multicentre longitudinal patient-reported outcomes study. BMC Med. 2021 Sep 28;19(1):227. doi: 10.1186/s12916-021-02098-y. PMID 34579718
- [Derived] Munyombwe T, Hall M, Dondo TB, Alabas OA, Gerard O, West RM, Pujades-Rodriguez M, Hall A, Gale CP. Quality of life trajectories in survivors of acute myocardial infarction: a national longitudinal study. Heart. 2020 Jan;106(1):33-39. doi: 10.1136/heartjnl-2019-315510. Epub 2019 Nov 7. PMID 31699696